CLINICAL TRIAL: NCT07133204
Title: Study of Efficacy and Safety of Cream Infused With HuangQin (Root of Scutellaria Baicalensis) Extract for the Reduction of Hyperpigmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mae Fah Luang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC 24061-25
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Hyperpigmentation; Melanin
Keywords: hyperpigmentation, scutellaria baicalensis, melanin index
MeSH Terms: conditions — Hyperpigmentation | interventions — Scutellaria baicalensis extract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental)
  Interventions: Other: Investigator developed cream infused with HuangQin extract

INTERVENTIONS:
Other: Investigator developed cream infused with HuangQin extract — A water in oil emulsion with consistency similar to cold cream. Infused with organic extract of scutellaria baicalensis.

SUMMARY:
The aim of this study is to evaluate the efficacy of a topical cream infused with Scutellaria baicalensis extract in reducing hyperpigmentation on the face.

The study is experimental clinical pilot study as a single group pretest-posttest.

A ROAT is conducted 1 week prior to the experiment. Participant apply the cream on the hypigmented area daily. Facial skin parameters (i.e. melanin index, erythema index) is evaluated at week 0, 1, 2 and 4.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Has at least 1 hyperpigmentation spot (size > 3mm) on either side of the face
* 30-60 y/o
* Fitzpatrick skin types II-IV
* Agrees to use sunscreen SPF50+ and willing to avoid strong sunlight exposure during the study

Exclusion Criteria:

* Pregnant or lactating
* Use of whitening products or treatment within 1 month before this study
* Currently using contraceptives
* History of allergy to any ingredient in the intervention cream
* Has skin conditions which can interfere with the measurement (i.e. severe acne, eczema, herpes simplex)
* Severe disease (i.e. immunodeficiency, cancer)
* Enrolled in other clinical study within 3 month before this study

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Efficacy of hyperpigmentation reduction property of the intervention | Week 0, 1, 2 and 4
  Measured the melanin index of the hyperpigmented area
Safefty profile of the intervention | Week 1, 2 and 4
  Record and collect the adverse effect from the usage of the interventional cream

SECONDARY OUTCOMES:
Efficacy of erythema reduction property of the intervention | Week 0, 1, 2 and 4
  Measured the erythema index of the hyperpigmented area
Efficacy of skin hydration property of the intervention | Week 0, 1, 2 and 4
  Measured the skin hydration value of the hyperpigmented area

CONTACTS AND LOCATIONS:
Overall Officials: Chakree C Wattanasiri, RPh PhD, Principal Investigator — Mae Fah Luang University
Locations (1):
- Mae Fah Luang University, Muang, Changwat Chiang Rai, Thailand

IPD SHARING:
Plan to Share IPD: No